CLINICAL TRIAL: NCT01341353
Title: Atrial Fibrillation Therapy: A Multi-Center Clinical Study
Brief Title: Catheter Ablation Versus Antiarrythmic Drugs for Atrial Fibrillation in China
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Collaborators: Capital Medical University (Other); Peking Union Medical College (Other); Guangdong Provincial People's Hospital (Other); Nanjing Medical University (Other); West China Hospital (Other); Dalian Medical University (Other); Shanghai Chest Hospital (Other)
Responsible Party: Cong-xin Huang,doctor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPA001
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Calcium Channel Blockers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiarrythmic Drugs (Active Comparator)
  Interventions: Drug: Digaoxin,amiodarone,β receptor antagonist, Calcium Antagonists
- ablation (Experimental)
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — circumferential pulmonary vein isolation complex fractionated atrial electrograms ablation circumferential pulmonary vein isolation combined left atrial roof ablation circumferential pulmonary vein isolation combined left atrial isthmus ablation circumferential pulmonary vein isolation combined left atrial roof and isthmus ablation circumferential pulmonary vein isolation combined complex fractionated atrial electrograms ablation
  Arms: ablation
Drug: Digaoxin,amiodarone,β receptor antagonist, Calcium Antagonists
  Arms: Antiarrythmic Drugs

SUMMARY:
The mainstay of treatment for atrial fibrillation remains pharmacological;however,catheter ablation has increasingly been used over the last decades. The relative merits of each strategy have not been extensively studied. Our study was designed to determine if catheter ablation is a feasible option as first-line therapy for treating patients with symptomatic AF.

ELIGIBILITY:
Inclusion Criteria:

* 1 Patients with symptomatic AF recorded by ECG or Holter 2 Age:18-75 years 3 Patients who are willing to enroll in the trial

Exclusion Criteria:

* 1 Patients accompanied hyperthyroidism 2 Patients with sever liver or renal dysfunction 3 Patients with sever cardiac dysfunction 4 Patients had previous radiofrequency catheter ablation in the LA or Maze surgical procedure 5 Patients with emboli in atrium 6 Pregnant woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with all-cause death | 3 month
Number of participants with all-cause death | 12 month
Number of participants with all-cause death | 24 month
Number of participants with all-cause death | 36 month
severe blooding complications | 3 month
severe blooding complications | 12 month
severe blooding complications | 24 month
severe blooding complications | 36 month
cardio-cerebrovascular complications | 3 month
cardio-cerebrovascular complications | 12 month
cardio-cerebrovascular complications | 24 month
cardio-cerebrovascular complications | 36 month
Number of participants with cardiovascular death events | 3 month
Number of participants with cardiovascular death events | 12 month
Number of participants with cardiovascular death events | 24 month
Number of participants with cardiovascular death events | 36 month

SECONDARY OUTCOMES:
recurrence of atrial arrhythmias (AF, AFL, AT) | 3 month
recurrence of atrial arrhythmias (AF, AFL, AT) | 12 month
recurrence of atrial arrhythmias (AF, AFL, AT) | 24 month
recurrence of atrial arrhythmias (AF, AFL, AT) | 36 month
resource utilization and costs | 12 month
resource utilization and costs | 24 month
resource utilization and costs | 36 month

CONTACTS AND LOCATIONS:
Overall Officials: Cong xin Huang, doctor, Study Chair — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China